CLINICAL TRIAL: NCT06258109
Title: Long-term Risk of Recurrent Cervical Artery Dissection After Pregnancy (LONG-RECAP Study)
Brief Title: Risk of Recurrent CeAD After Pregnancy
Acronym: LONG-RECAP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016_00547; ko23Engelter2
Record Dates: First submitted 2024-01-11; First posted 2024-02-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cervical Artery Dissection; Pregnancy Complications
Keywords: Ischemic Stroke; Hemorrhagic Stroke
MeSH Terms: conditions — Pregnancy Complications; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with pregnancy after index CeAD: Women who became pregnant at least once after first index CeAD
- Women without pregnancy after index CeAD: Women who did not became pregnant after first index CeAD

SUMMARY:
Primary objective: To determine whether pregnancy increases the risk of recurrent CeAD and delayed stroke in women with prior CeAD based on long-term data.

Methods: Multicentric, observational case-control study based on pooled individual patient data from several stroke centers.

Primary endpoint: Primary composite outcome measure includes the following outcomes: (i) occurrence of recurrent CeAD, (ii) occurrence of ischemic or hemorrhagic stroke, (iii) death.

DETAILED DESCRIPTION:
Background: Cervical artery dissection (CeAD) is a leading cause of stroke in women of childbearing age. Among the population with an initial CeAD, about 9% show a recurrence event (a range from 0 to 25% has been reported). Recurrence of CeAD can occur for several years after the initial event. CeAD has been shown to occur in association with pregnancy, and the postpartum period, yet it remains unclear whether pregnancy increases the risk of recurrence or delayed stroke. Previous studies on this subject are either based on small sample sizes or lack long-term data.

Objective: The investigators want to determine whether pregnancy increases the risk of recurrent CeAD and delayed stroke in women with prior CeAD based on long-term data.

Furthermore, it will be investigated whether the mode of delivery affects recurrence and if dissections occurred during a particular phase of a woman's reproductive process. The investigators will also investigate if women actively decided against another pregnancy due to the initial CeAD.

Methods: This study will be a multicenter, exploratory case-control study using pooled individual patient data from several stroke centers. The data will be obtained through review of medical records and patient interviews. The study will include all women with any prior CeAD who have had long-term follow-up (at least 6 months, with no upper limit), including information about pregnancy and recurrence of CeAD.

Primary endpoint is a composite outcome measure which consists of (i) occurrence of recurrent CeAD, (ii) occurrence of ischemic or hemorrhagic stroke, (iii) death. Secondary endpoints are the individual components of the primary endpoint and functional outcome assessed by the modified Ranking scale.

Statistical analysis will be used to determine the odds of the primary and secondary endpoints in women who had subsequent pregnancies compared to those who did not.

ELIGIBILITY:
Inclusion Criteria:

* female
* prior symptomatic cervical artery dissection (= index CeAD)
* at least one long-term follow-up visit (at least 6 months after the initial event)
* with information available on outcome events:
* recurrent dissection
* ischemic stroke
* hemorrhagic stroke
* functional outcome assessed by mRS score
* with data on pregnancy after the initial event
* at least 18 years old at the initial event

Exclusion Criteria:

* Male patients
* Age <18 years
* No long-term follow-up available or long-term follow-up < 6 months after initial event
* No data on pregnancy after initial event available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged ≥18 years with prior CeAD.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with composite outcome measure - recurrent CeAD, ischemic stroke, hemorrhagic stroke and/or death | From date of first CeAD until date of latest follow-up assessed up to 35 years
  The composite outcome measure includes the following outcome measures during the follow-up: (i) occurence of recurrent cervical artery dissection (CeAD), (ii) occurrence of any ischemic stroke, (iii) occurrence of any hemorrhagic stroke, (iv) death.

SECONDARY OUTCOMES:
Number of participants with recurrent cervical artery dissection | From date of first CeAD until date of latest follow-up assessed up to 35 years
  assessed by medical history or clinical suspicion with confirmation by cerebrovascular imaging (MRI, MRI angiography, CT, CT angiography, digital subtraction angiography and/or ultrasound)
Number of participants with new ischemic stroke | From date of first CeAD until date of latest follow-up assessed up to 35 years
  assessed by medical history or clinical suspicion with confirmation by cerebrovascular imaging (MRI and/or CT)
Number of participants with new hemorrhagic stroke | From date of first CeAD until date of latest follow-up assessed up to 35 years
  Intracerebral hemorrhage or subarachnoid hemorrhage assessed by medical history or clinical suspicion with confirmation by cerebrovascular imaging (MRI and/or CT)
Number of participants with death | From date of first CeAD until date of latest follow-up assessed up to 35 years
Functional outcome as assessed by modified Rankin Scale (mRS) | At date of latest, individual follow-up assessed up to 35 years after first CeAD
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan T Engelter, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (12):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Stroke Unit Sanatorio Allende, Córdoba, Argentina
- Department of Neurology, Medical University of Innsbruck, Innsbruck, Tyrol, Austria
- Helsinki University Central Hospital, Helsinki, Finland
- Germany (2):
  - Charité Universitätsmedizin, Centrum für Schlaganfallforschung, Berlin
  - Neurologische Klinik und Poliklinik, LMU Klinikum Campus Großhadern, Munich
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- Neurology Clinic, University of Brescia, Brescia, Italy
- Stroke Clinic, National Institute of Neurology and Neurosurgery Manuel Velasco Suárez, Mexico City, Mexico
- Switzerland (2):
  - University Hospital Basel, Stroke Center, Basel
  - University Hospital Zurich, Stroke Center, Zurich

IPD SHARING:
Plan to Share IPD: Undecided